CLINICAL TRIAL: NCT02531087
Title: Cross-Linked Collagen Peptides as a Urinary Biomarker of OI Pathobiology
Brief Title: Urinary Biomarkers of OI Pathobiology
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Shriners Hospitals for Children (Other); University of Nebraska (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Brendan Lee, Professor and Chairman, Baylor College of Medicine
Other Study IDs: 37358
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2024-12

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Individuals with OI: Individuals with OI with confirmed specific genetic mutations
- Controls/Unaffected: Individuals who do not have OI and who are not related to an individual with OI

SUMMARY:
Osteogenesis imperfecta (OI) is a rare inherited disorder that causes bones to break easily. Individuals with osteogenesis imperfecta break bones often and may have other problems, including hearing loss, dental problems, pain and difficulty getting around. Before the genetic cause of OI was known, OI was classified into four types. Each type was based upon the symptoms and severity of OI. In most people with OI, the cause is a change in one of the genes that makes a protein called type 1 collagen. Some doctors now classify OI both on how severe it is as well as which gene is causing OI. When people classify OI this way, there are more than 10 types of OI. The current laboratory testing to determine OI subtype involves the collection of blood and/or skin cells.

DETAILED DESCRIPTION:
Osteogenesis Imperfecta (OI) is a rare disorder that causes bones to break easily. People with OI may have broken bones with little or no trauma, dentinogenesis imperfecta (DI), and, in adult years, hearing loss. It is seen in both genders and all races. OI can range from very severe to very mild. Individuals with the most severe type of OI may die at birth. People with severe OI who survive may have bowed arms and legs, very short stature and be unable to walk. People with the mildest form of OI may only break bones occasionally and have normal height and lifespan. Breaks can occur in any bone, but are most common in the arms and legs. People with OI also often have problems with the spine. The spine problems include compression fractures and scoliosis (a curvature of the spine). DI is characterized by grey or brown teeth that may chip and wear down and break easily. In addition to weak teeth, the teeth in the upper jaw may not match up with the teeth in the lower jaw.

Before the genetic cause of OI was known, OI was classified into four types. Each type was based upon the symptoms and severity of OI. In most people with OI, the cause is a change in one of the genes that makes a protein called type 1 collagen. In the past decade, it was discovered that in about 5% of people with OI it is in another gene. Some doctors now classify OI both on how severe it is as well as which gene is causing OI. When people classify OI this way, there are more than 10 types of OI. The current laboratory testing to determine OI subtype involves the collection of blood and/or skin cells.

ELIGIBILITY:
Inclusion Criteria:

* To be able to participate, you must:

Be enrolled in The Longitudinal Study of OI (NTC #02432625) and have one of the following genetic mutations:

* glycine substitution mutations in COL1A1 or COL1A2
* haploinsufficient mutation in COL1A1 or COL1A2
* mutations in CRTAP, PPIB, or LEPRE1
* mutations in FKBP10 or SERPINH1
* mutations in (SERPINF1, WNT1, or IFITM5)
* dominant negative glycine substitutions and haploinsufficient mutations in COL1A1, and COL1A2

If you are serving as a control, you must not be related to an individual with OI.

Exclusion Criteria:

* You cannot participate if:
* You are unable to comply with the sample collection schedule.
* You are related to one of the OI subjects and would like to serve as a control subject.
* You have vertebral instrumentation or spinal deformities where we cannot assess lumbar spine aBMD.
* You have a history of recent fracture (< 3 months).
* You have serum creatinine above 1x upper limits of normal.
* You have abnormal kidney function.
* You are using Minoxidil.
* You are unable to provide a urine sample readily.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with OI
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
HP/LP Ratio | 5 Years
  The endpoint will be to compare the HP/LP ratio in OI patients with collagen overmodification (dominant negative mutations in COL1A1, COL1A2, and biallelic mutations in CRTAP, LEPRE1, PPIB) to those without overmodification (FKBP10, SERPINH1, IFITM5, SERPINF1, WNT1, and haploinsufficient mutations in COL1A1 and COL1A2).

SECONDARY OUTCOMES:
HP/LP ratio | 5 Years
  The endpoint would be the HP/LP ratio in those with dominant negative type I collagen mutations vs. those with mutations in P3H complex.

CONTACTS AND LOCATIONS:
Overall Officials: Vernon Reid Sutton, M.D., Principal Investigator — Baylor College of Medicine; Frank Rauch, M.D., Principal Investigator — Shriners Hospital for Children; David Eyre, Ph.D., Principal Investigator — University of Washington
Locations (7):
- United States (6):
  - University of California Los Angeles, Los Angeles, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Oregon Health Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Shriners Hospital for Children, Milwauke, Wisconsin
- Shriners Hospital for Children, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No